CLINICAL TRIAL: NCT02629107
Title: An All-Night Functional Magnetic Resonance Imaging Sleep Study With Auditory Stimuli
Brief Title: Functional Magnetic Resonance Imaging Sleep Study With Auditory Stimuli
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160031; 16-N-0031
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10-08

CONDITIONS: Normal Physiology
Keywords: Sleep; Functional Magnetic Resonance Imaging (fMRI); Electroencephalogram (EEG); Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy volunteers, age 18-34.

SUMMARY:
Background:

An electroencephalogram (EEG) measures the brain s electrical activity. EEG shows that the louder the sound needed to wake a person, the deeper the person s sleep. Researchers are using functional magnetic resonance imaging (fMRI) to study people during sleep so they can view brain activity in 3D. But they still need to correlate fMRI with sound thresholds, like the EEG.

Objective:

To measure brain activity during sleep using fMRI and EEG.

Eligibility:

Healthy people ages 18 34 who can sleep on their back for several hours.

Design:

Participants will be screened online about their sleep and general health.

At a screening visit, participants will have:

Physical exam

Hearing exam

MRI scan. A strong magnetic field and radio waves take pictures of the brain. Participants will lie down on a bed that slides into the scanner, which is shaped like a cylinder.

Participants will wear an actigraph on their wrist that records their motor activity.

Participants will follow a 2-week routine. This includes regular in-to-bed and out-of-bed times and limits on alcohol, caffeine, and nicotine.

During the overnight visits, participants will have:

Female subjects will have a urine pregnancy test.

fMRI. A coil will be placed over the head. Participants will do tasks shown on a computer screen inside the scanner.

EEG. Small electrodes on the scalp will record brain waves while sleeping or doing a task in the scanner.

Participants will be asked to try to sleep while researchers collect fMRI and EEG data. Participants eyes will be monitored with a video camera. Headphones will deliver sounds to wake them up throughout the night.

...

DETAILED DESCRIPTION:
Objective

Electroencephalography is generally considered the gold standard for defining sleep, but, in fact, sleep is a behavior and is defined by widely accepted behavioral characteristics like auditory arousal threshold. Electroencephalography merely became a surrogate for the behavioral definition when, in the first electroencephalographic sleep studies, researchers discovered a strong correlation between electroencephalographic slow waves and auditory arousal thresholds. With the advent of functional magnetic resonance imaging, one would expect the first sleep studies that used this new measure would have been designed to correlate it with auditory arousal threshold. However, these studies have never been conducted. This protocol will fill this gap in the literature. We hypothesize that undiscovered patterns of brain activity or functional connectivity exist during sleep and that an approach that defines sleep behaviorally will expose these patterns.

Study Population

The subject group in this study will be young, healthy individuals with excellent sleep health. Choosing this subject group will maximize the probability that subjects will sleep during all-night functional magnetic resonance imaging. Our target number of completers was 12 for the pilot study, was 43 for the main study, and is 85 for the normative study.

Design

After a one-week home-monitoring period that includes a regular in-to-bed and out-of-bed time, subjects will undergo two all-night functional magnetic resonance imaging sleep studies separated by a one-week washout period with continued home monitoring. The first night will serve as an adaptation night, which is known to reduce the sleep alterations that accompany sleeping in a laboratory environment. We will measure sleep depth behaviorally by arousing subjects with auditory stimuli that progressively increase in intensity. This procedure will be performed approximately eight times per night. The timing of the arousals will be distributed randomly across the night.

Data Generated

The data generated will be auditory arousal thresholds and the preceding brain activity and functional connectivity derived from functional magnetic resonance imaging.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. able to give informed consent;
  2. in good general heath;
  3. between the ages of 18 and 34 years;
  4. able to sleep on your back for several hours (with breaks).

EXCLUSION CRITERIA:

1. have a medical condition like diabetes or uncontrolled hypertension;
2. have a psychiatric or neurologic condition like depression or stroke;
3. have ever had a seizure;
4. have a sleep disorder like insomnia or sleep apnea;
5. work night shifts;
6. have metal in your body such as pacemakers, metal prostheses, or aneurysm clips that would make MRI scanning unsafe;
7. are pregnant or nursing;
8. drink too much caffeine (6 or more cups of coffee per day or 10 or more cups of caffeinated soda per day);
9. use too much alcohol (15 or more alcoholic beverages per week for men and 8 or more alcoholic beverages per week for women);
10. use too much nicotine (nicotine use within 30 minutes of waking);
11. are afraid of enclosed spaces;
12. have known hearing problems;
13. regularly use a prescription or over-the-counter drug to help you sleep or stay awake;
14. are an employee, contractor, or volunteer of the Laboratory of Functional and Molecular Imaging in the National Institute of Neurological Disorders and Stroke.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers will be recruited from the community and NIH employees.
Sampling Method: Non-Probability Sample
Enrollment: 2378 (Estimated)
Dates: Start 2016-01-14 (Actual); Primary Completion 2044-12-31 (Estimated); Study Completion 2045-12-31 (Estimated)

PRIMARY OUTCOMES:
The data generated will be auditory arousal thresholds and the preceding brain activity and functional connectivity derived from fMRI | This outcome will be measured during Overnight Visit 1 and 2.
  Auditory arousal thresholds will allow us to define sleep depth behaviorally.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Duyn, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moehlman TM, de Zwart JA, Chappel-Farley MG, Liu X, McClain IB, Chang C, Mandelkow H, Ozbay PS, Johnson NL, Bieber RE, Fernandez KA, King KA, Zalewski CK, Brewer CC, van Gelderen P, Duyn JH, Picchioni D. All-night functional magnetic resonance imaging sleep studies. J Neurosci Methods. 2019 Mar 15;316:83-98. doi: 10.1016/j.jneumeth.2018.09.019. Epub 2018 Sep 20. PMID 30243817
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-N-0031.html